CLINICAL TRIAL: NCT07319780
Title: A Multicenter Randomized Controlled Trial Comparing Fibrin-Enhanced Tubularized Incised Plate (F-TIP) and Grafted Tubularized Incised Plate (G-TIP) Urethroplasty in Distal Hypospadias With Unfavorable Urethral Plates
Brief Title: Fibrin-Enhanced TIP Versus Grafted TIP Urethroplasty in Distal Hypospadias
Acronym: FTIP-RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Children's Medical Center, Uzbekistan (Other)
Collaborators: Dr Cipto Mangunkusumo General Hospital (Other)
Responsible Party: Principal Investigator, Zafar Abdullaev, Head of the Pediatric Urology Department, National Children's Medical Center, Uzbekistan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 102025-11
Record Dates: First submitted 2025-12-20; First posted 2026-01-06 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Distal Hypospadias; Hypospadias
Keywords: Hypospadias repair; Tubularized incised plate; Platelet-rich fibrin; PRF; Grafted TIP; Pediatric urology
MeSH Terms: conditions — Hypospadias

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- F-TIP Urethroplasty (Experimental): Participants will undergo fibrin-enhanced tubularized incised plate (F-TIP) urethroplasty. Autologous platelet-rich fibrin will be prepared intraoperatively and applied to the incised urethral plate and fixed with PDS 6/0-7/0 suture prior to tubularization.
  Interventions: Procedure: Fibrin-Enhanced TIP Urethroplasty
- G-TIP Urethroplasty (Active Comparator): Participants will undergo grafted tubularized incised plate (G-TIP) urethroplasty using standard graft augmentation techniques for unfavorable urethral plates.
  Interventions: Procedure: Grafted TIP Urethroplasty

INTERVENTIONS:
Procedure: Fibrin-Enhanced TIP Urethroplasty — Tubularized incised plate urethroplasty augmented with autologous platelet-rich fibrin membrane applied to the incised urethral plate prior to tubularization.
  Arms: F-TIP Urethroplasty
Procedure: Grafted TIP Urethroplasty — Graft-augmented tubularized incised plate urethroplasty performed using standard surgical techniques for unfavorable urethral plates.
  Arms: G-TIP Urethroplasty

SUMMARY:
Hypospadias is a common congenital condition in boys in which the opening of the urethra is located on the underside of the penis. Distal hypospadias is the most common form and is usually treated surgically using tubularized incised plate (TIP) urethroplasty. In boys with an unfavorable urethral plate, graft-augmented techniques (G-TIP) are often used; however, postoperative complications such as urethrocutaneous fistula and narrowing of the urethral opening (meatal stenosis) may still occur.

Platelet-rich fibrin (PRF) is a biological material obtained from the patient's own blood that contains natural growth factors and may help improve tissue healing. This study aims to evaluate whether the use of PRF during surgery can reduce postoperative complications and improve surgical outcomes in children undergoing hypospadias repair.

DETAILED DESCRIPTION:
This is a prospective, multicenter, single-blinded randomized controlled trial designed to compare fibrin-enhanced tubularized incised plate (F-TIP) urethroplasty using autologous platelet-rich fibrin (PRF) with grafted tubularized incised plate (G-TIP) urethroplasty in children with distal hypospadias and an unfavorable urethral plate.

Male children aged 6 months to 84 months with primary or redo distal hypospadias and mild penile curvature will be eligible for inclusion. Participants will be randomized in a 1:1 ratio to undergo either F-TIP urethroplasty with intraoperative application of autologous PRF or standard G-TIP urethroplasty without PRF.

Autologous PRF will be prepared intraoperatively from the patient's peripheral blood using a standardized centrifugation protocol and applied to the incised urethral plate prior to tubularization.

Participants will be followed postoperatively for the assessment of surgical complications, functional outcomes, and cosmetic results according to predefined outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Male children aged 6 months to 84 months
* Primary or redo distal hypospadias
* Unfavorable urethral plate
* Penile curvature less than 45 degrees after degloving
* Eligibility for tubularized incised plate urethroplasty

Exclusion Criteria:

* Disorders of sex development or ambiguous genitalia
* Severe penile curvature requiring urethral plate transection
* Previous graft-based urethroplasty
* Active local or systemic infection at the time of surgery
* Known bleeding or platelet disorders
* Inability to comply with postoperative follow-up

Ages: 6 Months to 84 Months | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2026-01-05 (Actual); Primary Completion 2028-07-05 (Estimated); Study Completion 2028-12-25 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative urethral complications | 6 months postoperatively
  Incidence of postoperative urethral complications, defined as the occurrence of meatal stenosis requiring dilation or surgical intervention and/or urethrocutaneous fistula identified on clinical examination.

SECONDARY OUTCOMES:
Incidence of urethral stricture | 6 months postoperatively
  Presence of urethral stricture confirmed clinically or by imaging during follow-up.
Cosmetic outcome assessed by HOSE score | 6 months postoperatively
  Standardized postoperative photographs were assessed by two blinded external pediatric urologists using the Hypospadias Objective Scoring Evaluation (HOSE) system. HOSE scores range from 5 to 16 points, with higher scores indicating better cosmetic outcomes.
Maximum urinary flow rate (Qmax) | 6 months postoperatively
  Maximum urinary flow rate (Qmax), measured in milliliters per second (mL/s), assessed by uroflowmetry. Higher values indicate better urinary flow.

CONTACTS AND LOCATIONS:
Overall Officials: Zafar Abdullaev, MD, PhD, Principal Investigator — National Children's Medical Center, Tashkent, Uzbekistan
Locations (2):
- Dr. Cipto Mangunkusumo Hospital, Jakarta, DKI Jakarta, Indonesia
- National Children's Medical Center, Tashkent, Tashkent, Uzbekistan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Abbas TO, Khalil IA, Hatem M, Boyko A, Zorkin S. Plate Objective Scoring Tool (POST) in distal hypospadias: Correlation with post-repair complications. J Pediatr Urol. 2024 Apr;20(2):238.e1-238.e6. doi: 10.1016/j.jpurol.2023.11.022. Epub 2023 Nov 25. PMID 38071112
- [Result] Abbas TO. Evaluation of penile curvature in patients with hypospadias; gaps in the current practice and future perspectives. J Pediatr Urol. 2022 Apr;18(2):151-159. doi: 10.1016/j.jpurol.2021.12.015. Epub 2021 Dec 31. PMID 35031224
- [Result] Abbas TO. An objective hypospadias classification system. J Pediatr Urol. 2022 Aug;18(4):481.e1-481.e8. doi: 10.1016/j.jpurol.2022.05.001. Epub 2022 May 11. PMID 35644790